CLINICAL TRIAL: NCT05338463
Title: Evaluate the Safety and Efficacy of Fespixon Cream for the Treatment of Chronic Diabetic Foot Ulcers (TEXAS 1A, 2A) in Dialysis Patients
Brief Title: Fespixon Cream for the Treatment of Chronic Diabetic Foot Ulcers (TEXAS 1A, 2A) in Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cathay General Hospital (Other)
Collaborators: Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chi-Ming Pu, director of plastic surgery, Cathay General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ON101CLAS06
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Chronic Diabetic Foot Ulcer
Keywords: Chronic Diabetic Foot Ulcers (TEXAS 1A, 2A); Dialysis patients; Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Intervention Model Description: The study consists of 3 periods, a Screening/Run-in period, a treatment period, and a follow-up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fespixon Cream (Experimental): A single arm of Fespixon Cream for DFU (TEXAS 1A, 2A) in dialysis patients
  Test drug :
  1. Name : Fespixon Cream
  2. Dosage form: Topical cream, 15 g ointment per tube
  3. Active ingredients: 1.25% extracts of Plectranthus amboinicus (PA-F4, 0.25%) and Centella asiatica (S1, 1%)
  4. Dose(s): Apply 1 cc per 5 cm^2 ulcer size (not exceeding 2 mm in thickness)
  5. Dosing schedule: Apply twice a day
  6. Duration: up to 20 weeks
  Interventions: Drug: Fespixon Cream

INTERVENTIONS:
Drug: Fespixon Cream — 1. Name : Fespixon Cream
  2. Dosage form: Topical cream, 15 g ointment per tube
  3. Active ingredients: 1.25% extracts of Plectranthus amboinicus (PA-F4, 0.25%) and Centella asiatica (S1, 1%)
  4. Dose(s): Apply 1 cc per 5 cm^2 ulcer size (not exceeding 2 mm in thickness)
  5. Dosing schedule: Apply twice a day
  6. Duration: up to 20 weeks
  Other Names: ON101 Cream

SUMMARY:
Evaluate the Safety and Efficacy of Fespixon Cream for the Treatment of Chronic Diabetic Foot Ulcers (TEXAS 1A, 2A) in dialysis patients This study aimed to evaluate the effects of a topical cream containing Plectranthus amboinicus and Centella Asiatica when applied topically to diabetic foot ulcers in uremia patients with PAOD.

DETAILED DESCRIPTION:
This study is designed as a single-arm, open-label study to evaluate the efficacy and safety of Fespixon Cream for the treatment of chronic diabetic foot ulcers (DFUs) in dialysis.

Twelve(12) eligible subjects with DFUs and undergoing dialysis will be enrolled and assigned to receive Fespixon treatment for 20 weeks.

During the treatment phase, the Fespixon cream will be applied to the target ulcer twice a day for a maximum period of 20 weeks, until the ulcer closure (ulcer size of 0) for two consecutive visits at least 2 weeks apart, or until the subject exited the study as treatment failure. After that, all subjects regardless of wound healing at the end of the treatment phase will be followed for 2 weeks.

Identical standard of care (SoC) procedure will be performed throughout the study period, which including ulcer cleansing and debridement (if necessary) until complete ulcer closure.

At each visit, the size and changes of the target ulcer are recorded by photographing, and calculated using Image® software.

The study consists of three periods, a 2-week Screening/Run-in period, an up-to-20-week Treatment period, and a 2-week Follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, male or female, aged 20 to 80 years (inclusive) with Type 1 or Type 2 diabetes undergoing therapy for glycemic control using available diabetes drugs including insulin.
2. Subject has a glycosylated hemoglobin, HbA1c ≤ 12%.
3. Subjects maintain regular/stable blood purification treatment of hemodialysis (HD) or peritoneal dialysis (PD) for ≥6 months prior to Visit 0.
4. Presence of at least one diabetic foot ulcer that meets all of the following criteria:

   1. A full-thickness ulcer of UTWCS Grade I-A or II-A
   2. Ulcer size (area) is > 1 cm² and ≤ 10 cm² (post-debridement at time of enrollment)
   3. Ulcer is located on or below the malleoli.
   4. Ulcer presents for > 4 weeks (at time of enrollment).
   5. There is a minimum 3 cm margin between the qualifying Target Ulcer and any other ulcers on the specified foot, (post-debridement).
   6. No active infection by clinical inspection as defined by IDSA/IWGDF criteria. Note: If the subject has more than one qualifying diabetic foot ulcer, the most severe ulcer will be designated as the target ulcer; meanwhile, the depth of the wound will the consideration prior to the area of the wound.
5. Subject has adequate vascular perfusion of the affected limb, confirmed by Ankle-Brachial Index (ABI) ≥0.7 and < 1.3, transcutaneous pressure of oxygen (TcPO2) ≥30 mmHg on at least one lead, or Doppler ultrasound related test to ensure no serious embolisms/no serious clogging of blood vessels. .
6. Subject, if female of child-bearing potential, has a negative serum pregnancy test at screening, must not be breastfeeding, and willing to use 2 medically accepted methods of contraception (e.g., barrier contraceptives [female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectable, combination oral contraceptives, transdermal patches, or contraceptive rings], and intrauterine devices) during the course of the study (excluding women who are not of childbearing potential and/or who have been sterilized).
7. Subject is willing to use an off-loading device for the target ulcer on the plantar while ambulation for the duration of the study.
8. Subject / identified caregiver trained on the study procedures is able and willing to comply with study procedures.
9. A signed and dated informed consent form has been obtained from the subject prior to any study-related procedures being performed.

Exclusion Criteria:

1. In response to standard of care, ulcer size reduction is > 30% during the two-week run-in Screening Period (between the first Screening Visit/V0 and Baseline/V1).
2. Body mass index (BMI) > 35 kg/m2
3. Laboratory values at Screening of:

   1. Hemoglobin < 6.0 g/dL
   2. White Blood Cells (WBC) < 3.0 X 103 cells/uL； > 12.0 X 103 cells/uL
   3. Liver function studies [Total bilirubin, aspartate aminotransferase (AST) and alanine transaminase (ALT)] > 3x the upper limit of normal
   4. Albumin < 2.5 g/dL
4. Presence of any clinically significant medical condition(s) in medical history during screening period that, in the opinion of the investigator, could interfere with wound healing, including but not limited to the following:

   1. Acute or unstable Charcot foot
   2. Active malignant disease. A subject, who has had a malignant disease in the past, was treated and is currently disease-free, may be considered for study entry.
   3. Acquired immune deficiency syndrome (AIDS) or HIV positive.
5. Subject is currently receiving (i.e., within 30 days of enrollment visit) or scheduled to receive any of following medication or therapies, could interfere with wound healing during the course of the study.

   1. immunosuppressant (including chronic systemic corticosteroids)
   2. cytotoxic chemotherapy
   3. cytostatic therapy
   4. autoimmune disease therapy
   5. growth factors
   6. hyperbaric oxygen therapy
   7. bioengineered tissue or skin substitutes（ADM）
   8. application of topical steroids to the ulcer
   9. use of any investigational drug(s)
6. A psychiatric condition (e.g., suicidal ideation), current or chronic alcohol or drug abuse, determined from the subject's medical history, which, in the opinion of the investigator, may pose a threat to subject compliance.
7. Has any other factor which may, in the opinion of the investigator, compromise participation and/or follow-up in the study.

   Note ( Based on TEXAS 1A, 2A, the below information is to further calcification, and potential subjects meeting any of the following items will be excluded from the study.) :
   1. Ulcers with exposed bone or associated with osteomyelitis. (The osteomyelitis should be ruled out by clinical examination (probing of the wound) or X-ray findings as deemed necessary by the Investigator.)
   2. Presence of necrosis, purulence or sinus tracts that cannot be removed by debridement.
   3. Current sepsis
   4. Subjects who need to stand continuously for more than 4 hours / day and have difficulty complying with off-loading instructions.
8. The following products and ulcer care materials should NOT be used on or around the Target Ulcer after the first Screening Visit or at any time during the Treatment Phase of the study.

   1. Topical antibiotics, antiseptic soaps, steroids, or any other topical agents on the Target Ulcer.

      Note: Topical medication applied to the skin surrounding the Target Ulcer is allowed. (i.e. Skin barrier prep to protect peri-wound skin.)
   2. Hydrocolloid dressings are allowed only during the screening period but are not permitted after randomization.
   3. Hydrogelsare allowed only during the screening period but are not permitted after randomization.
   4. Silver nitrate hemostatic sticks or styptic pencils
   5. Negative pressure assisted closure device
   6. Heat lamps
   7. UV lights
   8. Whirlpool baths
   9. Water Piks
   10. Hyperbaric Oxygen
   11. Jet water streams (other than gentle saline irrigation) on the leg with Target Ulcer
   12. Ulcer dressings that include growth factors, engineered tissues or skin substitutes (e.g., Regranex®, Dermagraft®, Apligraf®, GraftJacket®, OASIS®, Primatrix®, Matristem®, etc.) on all ulcers including non-target ulcers during the Treatment Phase.
   13. Revascularization surgery on the leg with Target Ulcer
   14. Systemic steroids/oral corticosteroids (NOTE: inhaled steroids are acceptable)
   15. Other Immunosuppressive agents
   16. Autoimmune disease therapies
   17. Cytostatic drugs
   18. Any other investigational treatment/medications

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related Adverse Events associated with Fespixon cream | Time Frame: 20 weeks
  Assessment of Safety: Safety will be assessed based on the incidence of adverse events, including overall AEs, Fespixon-related AEs, target ulcer-related AEs, and SAEs.
  During the trial, in addition to self-reported AEs, physicians will check physical examination, vital signs, and laboratory reports to determine the presence of AEs

SECONDARY OUTCOMES:
Incidence of complete healing of the target ulcer | Time Frame: 20 weeks
  Incidence of complete healing of the target ulcer : measured by the photo to ensure the target ulcer area, such as length, width,and depth changed.
Time to complete ulcer healing | Time Frame: 20 weeks
  Time to complete ulcer healing : measured by the photo to ensure the target ulcer area, such as length, width,and depth changed.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Ming Pu, MD, Principal Investigator — Cathay General Hospital
Locations (1):
- Cathay General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
IIS study